CLINICAL TRIAL: NCT01927159
Title: A Phase 1b, Randomized, Double-blind, Placebo-controlled, Dose-escalation Study to Evaluate the Safety and Immunogenicity of the ID93 + GLA-SE Vaccine in BCG-Vaccinated Healthy Adults
Brief Title: Phase 1 ID93 + GLA-SE Vaccine Trial in BCG-Vaccinated Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Access to Advanced Health Institute (AAHI) (Other)
Collaborators: Aeras (Other); South African Tuberculosis Vaccine Initiative (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IDRI-TBVPX-114
Record Dates: First submitted 2013-08-15; First posted 2013-08-22 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Pulmonary Tuberculosis
Keywords: Tuberculosis; TB; Pulmonary; Vaccine; Adjuvant
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 10 mcg ID93 + 2 mcg GLA-SE Vaccine (QFT-) (Experimental): Three intramuscular injections of ID93 + GLA-SE at Days 0, 28, and 112. High dose of antigen and low dose of adjuvant. This group limited to adults with negative Quantiferon Gold TB (QFT) test.
  Interventions: Biological: ID93 + GLA-SE
- 2 mcg ID93 + 2 mcg GLA-SE Vaccine (Experimental): Three intramuscular injections of ID93 + GLA-SE at Days 0, 28, and 112. Low dose of antigen and low dose of adjuvant.
  Interventions: Biological: ID93 + GLA-SE
- 10 mcg ID93 + 2 mcg GLA-SE Vaccine (Experimental): Three intramuscular injections of ID93 + GLA-SE at Days 0, 28, and 112. High dose of antigen and low dose of adjuvant.
  Interventions: Biological: ID93 + GLA-SE
- 10 mcg ID93 + 5 mcg GLA-SE Vaccine (Experimental): Three intramuscular injections of ID93 + GLA-SE at Days 0, 28, and 112. High dose of antigen and high dose of adjuvant.
  Interventions: Biological: ID93 + GLA-SE
- Saline (Placebo Comparator): Three intramuscular injections of saline at Days 0, 28, and 112.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ID93 + GLA-SE
  Arms: 10 mcg ID93 + 2 mcg GLA-SE Vaccine; 10 mcg ID93 + 2 mcg GLA-SE Vaccine (QFT-); 10 mcg ID93 + 5 mcg GLA-SE Vaccine; 2 mcg ID93 + 2 mcg GLA-SE Vaccine
Other: Placebo
  Arms: Saline

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and immunogenicity in BCG-vaccinated healthy adult subjects of an investigational vaccine being developed for the prevention of pulmonary tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

1. Has completed the written informed consent process prior to start of screening evaluations
2. Male or female who is ≥18 years and ≤50 years of age at the time of randomization
3. Agrees to stay in contact with the study site for the duration of the study, provide updated contact information as necessary, and has no current plans to move from the study area for the duration of the study
4. Agrees to avoid elective surgery for the full duration of the study
5. For female participants: agrees to avoid pregnancy from 21 days prior to Study Day 0 and for the full duration of the study. Women physically capable of pregnancy (not sterilized and still menstruating or within 1 year of the last menses if menopausal) in sexual relationships with men must use an acceptable method of avoiding pregnancy during this period. Acceptable methods of avoiding pregnancy include a sterile sexual partner, sexual abstinence(not engaging in sexual intercourse), hormonal contraceptives (oral, injection, transdermal patch, or implant), vaginal ring, intrauterine device (IUD), or the combination of a condom or diaphragm with spermicide gel
6. Has general good health, confirmed by medical history and physical examination
7. Has body mass index (BMI) between 19 and 33 (weight/height2) by nomogram
8. Had BCG vaccination at least 5 years ago, documented through medical history or presence of scar

Exclusion Criteria:

1. Acute illness at the time of randomization
2. Oral temperature ≥37.5°C at the time of randomization
3. Clinically significant abnormal laboratory values for any of the following screening laboratory parameters, per local laboratory normal ranges from blood collected within 30 days prior to Study Day 0 randomization as follows:

   * hemoglobin, hematocrit, absolute neutrophil count, absolute lymphocyte count, or platelet count below lower limit of normal (LLN)
   * white blood cell count above upper limit of normal (ULN) or below LLN (i.e., must be within normal limits)
   * ALT, AST, total bilirubin, alkaline phosphatase, creatinine, or blood urea nitrogen (BUN) above ULN
4. Evidence of systemic or local disease process on screening urinalysis
5. Evidence of significant active infection
6. History of treatment for active or latent tuberculosis or evidence of active tuberculosis
7. Shared a residence within the last year prior to randomization with an individual on anti-tuberculosis treatment or with culture or smear positive tuberculosis
8. History of autoimmune disease or immunosuppression
9. Used immunosuppressive medication within 42 days before randomization (inhaled and topical corticosteroids are permitted)
10. Received immunoglobulin or blood products within 42 days before randomization
11. Received any investigational drug therapy or investigational vaccine within 182 days before randomization, or planned participation in any other investigational study during the study period
12. Received investigational Mtb vaccine at any time prior to randomization
13. Received a live vaccine within past 4 weeks or a killed vaccine within past 2 weeks prior to randomization.
14. Unable to discontinue current chronic prescription drug therapy that can be hepatotoxic or toxic to the bone marrow or kidneys.
15. History or laboratory evidence of immunodeficiency state including but not limited to any laboratory indication of HIV-1 infection
16. History of allergic disease or reactions (including allergy to kanamycin-related antibiotics, allergic reaction to eggs, and severe eczema), likely to be exacerbated by any component of the study vaccine
17. Previous medical history that may compromise the safety of the participant in the study, including but not limited to: severe impairment of pulmonary function from pulmonary disease; chronic illness with signs of cardiac or renal failure; suspected progressive neurological disease; or uncontrolled epilepsy
18. Evidence of chronic hepatitis (e.g., hepatitis B surface antigen or hepatitis C antibody)
19. Chronic heavy ethanol intake which, in the opinion of the investigator, may compromise the safety of the participant or interfere with the evaluation of the safety of the vaccine
20. Cannabis smoking 3 or more days per week
21. Positive urine test for illicit drugs (opiates, cocaine, amphetamines)
22. History or evidence on physical examination of any systemic disease or any acute or chronic illness that, in the opinion of the investigator, may interfere with the evaluation of the safety or immunogenicity of the vaccine
23. All female participants: currently pregnant or lactating/nursing; or positive urine pregnancy test during screening or on the day of study injection
24. Received a tuberculin skin test within 3 months (90 days) prior to Study Day 0
25. Any current medical, psychiatric, occupational, or substance abuse problems that, in the opinion of the investigator, will make it unlikely that the participant will comply with the protocol or may compromise the safety of the participant

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2013-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 294 days
  Solicited and unsolicited adverse events will be recorded for 28 days following each study injection; serious adverse events and adverse events of special interest will be recorded for the duration of the study.

SECONDARY OUTCOMES:
Immunogenicity | Days 0, 14, 42, 112, 126, 196, 294
  Immunogenicity will be evaluated by measuring humoral and cellular responses to ID93 + GLA-SE at specified timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Tameris, M.B.Ch.B., Principal Investigator — SATVI
Locations (1):
- SATVI, Worcester, Western Cape, South Africa

REFERENCES:
- [Derived] Penn-Nicholson A, Tameris M, Smit E, Day TA, Musvosvi M, Jayashankar L, Vergara J, Mabwe S, Bilek N, Geldenhuys H, Luabeya AK, Ellis R, Ginsberg AM, Hanekom WA, Reed SG, Coler RN, Scriba TJ, Hatherill M; TBVPX-114 study team. Safety and immunogenicity of the novel tuberculosis vaccine ID93 + GLA-SE in BCG-vaccinated healthy adults in South Africa: a randomised, double-blind, placebo-controlled phase 1 trial. Lancet Respir Med. 2018 Apr;6(4):287-298. doi: 10.1016/S2213-2600(18)30077-8. PMID 29595510

DOCUMENTS (1):
  • Study Protocol (2013-02-08): https://cdn.clinicaltrials.gov/large-docs/59/NCT01927159/Prot_000.pdf